CLINICAL TRIAL: NCT00175708
Title: Pedobarographic Assessments of Clubfoot Treated Patients
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christine Alvarez, Principle Investigator, University of British Columbia
Other Study IDs: H03-70531
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2017-05

CONDITIONS: Clubfoot
Keywords: Evaluation of an outcome tool; clubfoot; foot pressure profiles; pedobarographs
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the utility of pedobarographs in evaluating clubfoot post-treatment.

DETAILED DESCRIPTION:
Detailed Description: Using Tekscan's HRMat Pressure assessment system or EMED pedobarography system the distribution of force will be measured across the plantar surface of the subject' foot. The Tekscan system is comprised of a 50 cm square pressure sensor connected to a computer interface. The data collection will be made up of two parts:

Part I: Static Profile: The child will be asked to stand on the mat for 6 seconds for five trials. During this time the data collection software will collect force data across the foot 60 times per second. The software will then calculate centre of force as well as changes in pressure during the static trial. The foot will be assessed into the distribution of forces across the hindfoot, midfoot, forefoot, and the big toe. In addition, the centre of gravity will also be determined.

Part II: Dynamic Profile: The dynamic test will involve the child walking across the mat for a total of 5 passes per foot. Measurements of force will again be taken at 60 Hz.

The EMED-x400 sensor is rectangular and its dimensions are 47.5 cm by 32 cm. Measurements of force will be recorded at up to rates of 400 Hz. Foam pieces (included with the EMED platform) are constructed around the platform to establish a levelled and safe runway for the patient to walk along. The EMED platform is connected to a computer interface which operates on the Novel analysis software. The subject will be asked to walk across the mat independently at their ordinary pace. The foot is required to land in the centre of the mat, at a minimum of three trials per foot10. Plantar pressure recording takes 10-20 minutes for each subject.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria - all clubfoot patients seen at BC Children's Hospital who have commenced walking and compliant to the study protocol. As the goal of the study is to evaluate the utility of pedobarographs in evaluating clubfoot treatment, we will be following subjects with all presentations of clubfoot (this includes idiopathic clubfoot and clubfoot that is secondary to another global disorder).

Exclusion Criteria:

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Clubfoot patients seen at BC Children's Hospital in Vancouver.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2005-09; Primary Completion 2016-06 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christine Alvarez, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Department of Orthopaedics, Vancouver, British Columbia, Canada